CLINICAL TRIAL: NCT03785093
Title: Intestinal Microbiota on Allergy, Growth and Development of the Next Generation in Hong Kong
Brief Title: Intestinal Microbiota on Allergy, Growth and Development
Acronym: SMARTGenHK
Status: Active, not recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ting-fan Leung, Professor, Chinese University of Hong Kong
Other Study IDs: Smart-002
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Pregnancy
Keywords: Microbiota, Allergy, Growth, Development, offspring
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — i) Blood, urine and stool samples ii) Skin, nasal and buccal swabs iii) Maternal vaginal swabs and placental tissue biopsy iv) Breast milk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chinese Family: Chinese parents and their offsprings

SUMMARY:
There is growing evidence that microbial programming beginning in-utero can be a central component for a balanced development of innate immunity and optimal growth and development in newborns. However, the specific types of bacteria along with their cross-talk with maternal and fetal host factors are far from being clear. The investigators hypothesize microbial compositions at different body sites of pregnant women are associated with early-life microbiota of their offspring as well as growth, neurodevelopment and the development of allergic and neurocognitive disorders. This is a prospective birth cohort study involving Chinese mother-child pairs. The investigators will follow up 120 pregnant women from first trimester until childbirth, and the child until three years of age.

DETAILED DESCRIPTION:
Our unit is one of the centres contributing to the International multicentre HAPO study. We recruited 1760 Chinese pregnant women between 2000 and 2005. The HAPO study investigated whether any adverse outcome was associated with mild degree of GDM. All mothers underwent a 75-gram OGTT at 24-32 weeks gestation, but clinicians were blinded to the results as long as the fasting PG was ≤ 5.8 mmol/L & 2-hour PG ≤ 11.1 mmol/L. The maternal serum C-peptide and HbA1c, cord serum C-peptide and early neonatal PG, pregnancy outcome and the neonatal anthropometric parameters are available for future study. This is so far the largest cohort in a Chinese population who has been investigated for glycaemia during pregnancy, but with OGTT results remained undisclosed to subjects and clinicians. This unique cohort can allow us to study the effect of in-utero hyperglycemia on the cardiometabolic risks at childhood, adolescence and adulthood.

Eligible subjects are all mother-child pairs participating in the original HAPO study. Children born preterm before 37 weeks of gestation, non-Chinese and whose mother's OGTT result were unblinded during pregnancy will be excluded.The family (the child and the mother) will be invited for a third follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Expectant ethnic Chinese mothers aged 18 - 45 years who are in the first trimester of pregnancy
2. Singleton pregnancy
3. Plan to give birth in the Prince of Wales Hospital, Hong Kong and stay with the child in Hong Kong for the next 3 years
4. Willing to provide serial biological samples for microbiota detection
5. Willing for her coming newborn to be prospectively followed up for clinical and microbiota data collection in PWH
6. Participate voluntarily and capable of giving informed consent

Exclusion Criteria:

1. Significant medical conditions especially those required long term medications, such as oral steroid, antihypertensive drugs, diabetic medications and lipid-lowering agents, during or before pregnancy
2. History of chronic inflammatory or neoplastic diseases involving the gastrointestinal tract (e.g. inflammatory bowel disease, coeliac disease, colorectal cancer)
3. Significant pregnancy complications, such as intrauterine foetal demise/stillbirth, extreme prematurity, or pre-labour rupture of membranes before 24 weeks
4. Mother with mental incapacity such that they are not able to give informed consent
5. Foetal chromosomal or clinically significant structural abnormalities
6. The current pregnancy is a conception through either sperm or ovum donation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women who are in the first trimester of pregnancy
Study Population: Chinese families in Hong Kong
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Composite allergy disease | 3 years of age
  wheezing, asthma, skin atopy, food allergy

CONTACTS AND LOCATIONS:
Overall Officials: Ting Fan Leung, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong, China, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] He Y, Zhang L, Chen Z, Chan PKS, Leung TF, Tam WH. The associations of pre-pregnancy BMI and gestational weight gain with maternal gut microbiota. Benef Microbes. 2024 Jul 3;15(4):397-410. doi: 10.1163/18762891-bja00018. PMID 38955351